CLINICAL TRIAL: NCT06064513
Title: The Effect of Video-Based Empathy Training on Empathy Skills and Integrative Nursing Competence Level in Nurses-Randomized Controlled Study
Brief Title: Video-Based Empathy Training for Nurses
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, Cevriye Ozdemir, Phd RN Assistant Professor, Saglik Bilimleri Universitesi
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: SY200217B07
Record Dates: First submitted 2023-09-26; First posted 2023-10-03 (Actual); Last update posted 2023-10-03 (Actual); Status verified 2023-09

CONDITIONS: Empathy; Humanism
Keywords: Empathy; Nursing; Wholistic Health Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (Experimental): It consists of nurses working in Intensive Care, Emergency Service, Internal - Surgical Services and Polyclinic units in the public hospital in Kayseri. Individuals who volunteer to participate in the research will be included.
  Interventions: Other: verbal empathy training
- Video group (Experimental): It consists of nurses working in Intensive Care, Emergency Service, Internal - Surgical Services and Polyclinic units in the public hospital in Kayseri. Individuals who volunteer to participate in the research will be included.
  Interventions: Other: video based empathy training

INTERVENTIONS:
Other: verbal empathy training — Empathy training will be given to nurses in the control group using face-to-face interview technique. In this training, the researcher will explain verbally what empathy is and how to make an empathetic approach to sick individuals. The training will be given to nurses twice, one week apart, at their own time.
  Arms: control group
Other: video based empathy training — Nurses in the video group will be shown a video recording about empathy. Nurses will be allowed to watch the training video twice, with an interval of one week. After the empathy training is completed, the evaluation phase will begin. For this purpose, 2 weeks and 4 weeks after the end of the last training, nurses in both study groups will be asked to fill out the Integrative Nursing Competency Scale and Empathy Level Determination Scale. In the study, a comparison of nurses' pre-test and post-test answers will be made to evaluate the effectiveness of video-based education.
  Arms: Video group

SUMMARY:
Nurses should provide health care services to healthy/sick individuals, families and society with a holistic and holistic approach. Nurses, who are holistic care providers, see the individual/patient as a whole within his own environment and know that he consists of body, mind and spirit. In general, holistic care addresses people's physical, mental, emotional and spiritual needs, enabling them to cope with their illnesses and improve their lives. The helpful and supportive nature of the nursing profession is always at the forefront. Empathy in nursing care is one of the basic components of the relationship established with the nurse and the person being cared for. In a holistic and humanistic approach, nurses need to approach individuals with an empathetic attitude in order to understand their needs correctly and achieve more positive results. However, the nursing profession has difficulty in establishing empathy due to many negative factors in the work environment and cannot exhibit a humanistic approach. Based on this, it was aimed to determine the effect of video-based empathy training on nurses' empathy skill level and holistic nursing competence.

DETAILED DESCRIPTION:
This study was designed as a randomized controlled study to determine the effect of video-based empathy training on the empathy skill level and holistic nursing competence level of nurses. The population of the research will consist of nurses working in two public hospitals in Kayseri. In this study, G-Power power analysis program was used to determine the number of samples. Using the Cohen standardized effect size for the study, the minimum sample size was calculated as 34 for each group, with a medium effect size (0.5), alpha value of 5%, and theoretical power of 80%. The importance of increasing the sample size to control bias due to losses and the acceptability of data loss below 10%-15% are emphasized. For this reason, 15% more individuals will be included in the study and 80 nurses will be included in the study. Descriptive characteristics information form, holistic nursing competency scale, and empathy level determination scale will be used to collect research data. Empathy Training Video: The empathy-themed video that will be used within the scope of the research belongs to Cleveland Clinic. Permission for use was obtained after contacting the institution via e-mail and providing information about the research. The video is in Turkish and translated by the institution. Cleveland Clinic is a nonprofit American academic medical center based in Ohio. In the video content, language, religion, race, age, gender, etc. The importance of taking an empathetic approach to individuals regardless of their needs is explained. Patients included in the study will be divided into two groups: control and video groups. Participants in both groups will be asked to fill out an introductory characteristics information form, holistic nursing competency scale, and empathy level determination scale. Empathy training will be given to nurses in the control group using face-to-face interview technique. In this training, the researcher will explain verbally what empathy is and how to make an empathetic approach to sick individuals. The training will be given to nurses twice, one week apart, at their own time. Nurses in the video group will be shown a video recording about empathy. Nurses will be allowed to watch the training video twice, with an interval of one week. After the empathy training is completed, the evaluation phase will begin. For this purpose, 2 weeks and 4 weeks after the end of the last training, nurses in both study groups will be asked to fill out the Integrative Nursing Competency Scale and Empathy Level Determination Scale. In the study, nurses' pre-test and post-test answers will be compared to evaluate the effectiveness of video-based education. The data obtained from the study will be evaluated in the IBM SPSS 24 Statistics (Statistical Package for the Social Sciences) package program.

ELIGIBILITY:
Inclusion Criteria:

* Being a nurse working in a public hospital in Kayseri,
* Being a nurse working in intensive care, emergency service, internal - surgical services and polyclinic units,
* Individuals who volunteer to participate in the research will be included.

Exclusion Criteria:

* Being a nurse working outside the specified services,

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-10-01 (Estimated); Primary Completion 2023-10-15 (Estimated); Study Completion 2023-12-15 (Estimated)

PRIMARY OUTCOMES:
Integrative Nursing Competence | 2 months
  They will be asked to complete the Integrative Nursing Competency Scale.

SECONDARY OUTCOMES:
Empathy Level | 2 months
  They will be asked to fill out the Empathy Level Determination Scale.

CONTACTS AND LOCATIONS:
Overall Officials: Cevriye Ozdemir, PhD RN, Principal Investigator — Saglik Bilimleri University
Locations (1):
- Saglik Bilimleri University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Information about the research can be obtained at any time by contacting the authors.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: It can be obtained within 6 months after the research is published.
Access Criteria: Becoming a researcher in the field of nursing